CLINICAL TRIAL: NCT00334503
Title: Open Trial of Miglitol in Type 2 Diabetic Patients Treated With Biguanide
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG1009
Record Dates: First submitted 2006-06-05; First posted 2006-06-07 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: alpa-glucosidase inhibitor,Biguanide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — miglitol

INTERVENTIONS:
Drug: Miglitol

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy and safety of Miglitol in patients with Type2 Diabetes Mellitus treated with Biguanide.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetic patients with Biguanide treatment
* Criteria for postprandial plasma glucose and HbA1c are met

Exclusion Criteria:

* Type 1 diabetes
* Patients treated with other antidiabetic drugs or Insulin

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Group, Clinical Development Dept., Study Director — Sanwa Kagaku Kenkyusho Co., Ltd.
Locations (13):
- Japan (13):
  - Aichi
  - Chiba
  - Fukuoka
  - Gunma
  - Hokkaido
  - Ibaraki
  - Kagoshima
  - Kanagawa
  - Kumamoto
  - Miyazaki
  - Osaka
  - Ōita
  - Saitama